CLINICAL TRIAL: NCT02458404
Title: Effects of Varied Estrogen Doses on Endometrial Receptivity
Status: Completed | Type: Observational
Sponsor: Reproductive Medicine Associates of New Jersey (Other)
Responsible Party: Sponsor
Other Study IDs: RMA-2014-03
Record Dates: First submitted 2015-03-31; First posted 2015-06-01 (Estimated); Last update posted 2019-11-07 (Actual); Status verified 2019-11

CONDITIONS: Luteal Phase Defect

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This study will help determine the effect of varied estradiol levels on the uterine lining in healthy humans that are not undergoing a stimulated in vitro fertilization (IVF) cycle.

DETAILED DESCRIPTION:
Volunteers who wish to participate in the study, will undergo a diagnostic and screening phase to determine their eligibility. Once eligibility is determined, participants will undergo three, separate "endometrial preparatory cycles". These cycles will consist of estrogen supplementation to mimic normal, above normal, and highly elevated estradiol levels. Once supplementation is complete uterine procedures will be done to hopefully determine the effects of the estrogen levels on the uterine lining. Subcutaneous leuprolide injections, intramuscular estrogen, and progesterone injections will be used to mimic the levels needed. Blood draws will monitor the needed estradiol and progesterone levels during the injection phase of the cycle. Once the injection phase is complete, transvaginal ultrasound, uterine aspiration, and endometrial biopsy will be done.

ELIGIBILITY:
Inclusion Criteria:

* Regular menstrual cycles
* Age 18-50
* Normal Baseline ultrasound
* No intra-uterine procedures in prior 90 days

Exclusion Criteria:

* Any contraindications to undergoing estrogen stimulation of the endometrium
* Age ≥35 years and smoking ≥15 cigarettes per day
* Multiple risk factors for arterial cardiovascular disease (smoking, diabetes, and hypertension)
* Hypertension (systolic ≥140 mmHg or diastolic ≥90 mmHg)
* Venous thromboembolism (current or history of)
* Known thrombogenic mutations
* Known ischemic heart disease
* History of stroke
* Complicated valvular heart disease (pulmonary hypertension, risk for atrial fibrillation, history of subacute bacterial endocarditis)
* Systemic lupus erythematosus (positive or unknown antiphospholipid antibodies)
* Migraine with aura at any age
* Breast cancer
* Cirrhosis
* Hepatocellular adenoma or malignant hepatoma
* History of undiagnosed abnormal uterine bleeding.
* Allergic reaction to any study drug
* Known pregnancy or delivery within the past 6 months
* Breastfeeding
* Obesity >35 kg/m2

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy human subjects
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2015-03 (Actual); Primary Completion 2017-01 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Endometrial thickness in millimeters as assessed by transvaginal ultrasound | Participants will be followed for the duration of 1 menstrual cycle, ~30 days; this is followed by 1 rest mentrual cycle, ~30 days; there are a total of 3 rest and 3 treatment cycles, ~180 days
  1. Participants will undergo 3 transvaginal ultrasounds. Endometrial thickness will be recorded.
  2. Purpose: The serum hormone levels serve as the immunoassays while the endometrial lining serves as the bioassay. This will allow for baseline evaluation of the uterine lining and myometrium as well as monitor biological response to the estrogen and progesterone.
mRNA and protein expression of known markers of secretory transformation as assessed by real time PCR and immunohistochemistry after uterine aspiration and disruption/biops | Participants will be followed for the duration of 1 menstrual cycle, ~30 days; this is followed by 1 rest mentrual cycle, ~30 days; there are a total of 3 rest and 3 treatment cycles, ~180 days
  Patients will undergo a uterine aspiration and endometrial disruption/biopsy. These will be analyzed for known markers involved in human reproduction utilizing established molecular biological assessment tools. In particular markers which will be evaluated will be: LIF, CXCL13, beta 2 integrin, DAF, OPN, and IL15
Endometrial echotexture as assessed by transvaginal ultrasound | Participants will be followed for the duration of 1 menstrual cycle, ~30 days; this is followed by 1 rest mentrual cycle, ~30 days; there are a total of 3 rest and 3 treatment cycles, ~180 days
  a. Participants will undergo 3 transvaginal ultrasounds. Endometrial echotexture will be recorded.

SECONDARY OUTCOMES:
Peak and trough estrogen and progesterone levels as assessed by peripheral phlebotomy | Participants will be followed for the duration of 1 menstrual cycle, ~30 days; this is followed by 1 rest mentrual cycle, ~30 days; there are a total of 3 rest and 3 treatment cycles, ~180 days
  Peripheral phlebotomy will be performed in order to determine peak and trough levels of hormones.
Uterine microbiome characterization by microbiota presence and prevalence as assessed after uterine aspiration | Participants will be followed for the duration of 1 menstrual cycle, ~30 days; this is followed by 1 rest mentrual cycle, ~30 days; there are a total of 3 rest and 3 treatment cycles, ~180 days
  Patients will undergo a uterine aspiration. The human microbiome project has revealed important things about the vaginal microbiome, but little is known about the uterine microbiome. Given the hormonal changes change the pH of the vagina, we will be able to characterize differences in the uterine microbiome with varied estrogen levels.

CONTACTS AND LOCATIONS:
Overall Officials: Richard T Scott, MD, HCLD, Principal Investigator — RMA of NJ
Locations (1):
- Reproductive Medicine Associates of New Jersey, Basking Ridge, New Jersey, United States

REFERENCES:
- [Derived] Osman EK, Wang T, Zhan Y, Juneau CR, Morin SJ, Seli E, Scott RT, Franasiak JM. Varying levels of serum estradiol do not alter the timing of the early endometrial secretory transformation. Hum Reprod. 2020 Jul 1;35(7):1637-1647. doi: 10.1093/humrep/deaa135. PMID 32613240